CLINICAL TRIAL: NCT05839288
Title: Pyrotinib Plus Trastuzumab and Chemotherapy in Metastatic HER2-positive Breast Cancer Patients- a Multicenter Retrospective Study
Brief Title: Pyrotinib Plus Trastuzumab and Chemotherapy in HER2+ Metastatic Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-26
Record Dates: First submitted 2023-04-03; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
Keywords: Pyrotinib
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PyroHC: Patients used pyrotinib (Pyro) plus trastuzumab (H) and chemotherapy (C) as treatment for metastatic breast cancer.

SUMMARY:
To evaluate the patterns and treatment outcomes of pyrotinib plus trastuzumab and chemotherapy in the real world.

ELIGIBILITY:
Inclusion Criteria:

* woman, age > 18 years old
* diagnosed with HER2 +Metastatic Breast Cancer
* received pyrotinib plus trastuzumab and chemotherapy for at least one cycle, starting from 2018.07-2022.09
* available medical history

Exclusion Criteria:

* medical history was incomplete

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer (according to International Classification of Diseases-10, ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 6 weeks
  Progression free survival

SECONDARY OUTCOMES:
Adverse events | 6 weeks
  Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] You S, Sang D, Xu F, Luo T, Yuan P, Xie Y, Wang B. Real-world data of triplet combination of pyrotinib, trastuzumab, and chemotherapy in HER2-positive metastatic breast cancer: a multicenter, retrospective study. Ther Adv Med Oncol. 2023 Dec 23;15:17588359231217972. doi: 10.1177/17588359231217972. eCollection 2023. PMID 38145113